CLINICAL TRIAL: NCT02920138
Title: The Effect of PEEP, Zero PEEP and Intraabdominal Pressure Levels on Cerebral Oxygenation (rso2) in the Morbidly Obese Undergoing Sleeve Gastrectomy
Brief Title: The Effect of PEEP and Intraabdominal Pressure Levels on Cerebral Oxygenation Morbidly Obese.
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: DuzceU
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Unspecified Effect of Air Pressure
Keywords: Obesity; intraabdominal pressure; cerebral oxymeter; sleeve gastrectomy; laparoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 5PEEP: Administered 5 cmH2O positive end expiratory pressure group( Group 5PEEP n=30).
- Group ZEEP: no positive end expiratory pressure group (Group ZEEP n=30)

SUMMARY:
Background: Study was designed to determine the effect of zero (ZEEP) and 5 mmHg positive end expiratory pressure (5PEEP) on cerebral oximeter levels in morbid obese patients whose undergoing laparoscopic sleeve gastrectomy. Second outcome is to investigate the effect of intraabdominal pressure changes on cerebral oxygen values in LSG.

Method:18-65 yo, ASA2-3 status, 60 morbid obese patients which planned SLG under general anesthesia were included.Two patient in Group 5 PEEP were excluded because of the haemodynamic instability during procedure. Patients were divided into 2 groups which was ventilated with no PEEP (Group ZEEP)(n=30) and 5 cmH2O PEEP levels (Group5 PEEP)(n=28). All patients were use right hand dominant. Near infrared spectroscopy probes were applied to both frontal cerebral area of all patiens and measured rSO2 values. IAP were measured transvesically in all groups. Datas were recorded as basal, after induction of anesthesia, 5 minute before insufflation(5BI), 5 minute after insufflation(5BA), 15, 30, 45, 60 minute after induction, 5 minute before desufflation(5BD) and 5 minute after desufflation(5AD) time periods. Invasive arterial pressures, cerebral oxymeter values, 5 lead electrocardiography, peripheral oxygen saturation, end tidal carbondioxide, peak inspiratory pressures, intra abdominal pressure, were recorded time periods in all groups. Arterial blood sample analysed on 5BI,5AI, 5AD periods.

DETAILED DESCRIPTION:
60 morbidly obese patients which planned sleeve gastrectomy procedures under general anestesia (ASA 2-3 status) were included in this study. Patients were devided into 2 groups which was ventilated with no positive end expiratory pressure (Group 5PEEP n=30), and 5 cmH2O positive and expiratory pressure (Group ZEEP n=30). All the patients were right hand dominate.Two patient in Group 5 PEEP were excluded because of the haemodynamic instability during procedure.

Exclusion criteria: Documented coronary or periferally arteryel disease, unregulated diabetes mellitus, history of smoking, symptoms of bowel or urinary bladder obstruction, preoperative systolic pressure grater than 170 mmHg, diastolic arterial pressure grater than 90mmHg, pregnancy, anemia (haematocrit levels under %30), and symptoms of increased intracranial pressure, significant stenosis of the carotid arteries. In all anesthetised patients were monitorised with 3 leads electrocardiography(ECG), pulse oxymetry (sPO2),invasive blood pressure(IBP), end-tidal carbondioxide (EtCO2),intraabdominal pressure levels (IAP)with intravesical urinary catheter, peak inspiratuar pressure (PIP), laparoscopic pressure (LP), regional cerebral oxygen saturation(rSO2) continuously. rSO2 values were measured with near infrared spectroscopy (NIRS) technique by cerebral oximeter (INVOS 4100, Somanetics, Covidien) measurements recorded as basal values; after induction; before 15 minute of insufflation; after 15 minute of insufflation; 30, 45, 60 after induction; before 15 minute of desufflation; after 15 minute of desufflation. Arterial blood samples were collected and performed before 15 minute of insufflation; after 15 minute of insufflation; after 15 minute of desufflation. Partial oxygen pressure(PaO2), partial carbondioxide pressure( PaCO2), peripheric oxygen saturation (SaO2), bicarbonate (HCO3), aside- base status (pH), haematocrit (Htc) haemoglobin(Hb) levels were recorded and evaluated those three time periods which explained above. Cerebral oximeter was placed skin of the patients forehead after clean special skin-prep pad. The skin sensors were applied on the right and left sides of the forehead. The medial margin of the sensor was at the midline of the forehead and lateral margin 2 cm above the eyebrows.

After induction of anesthesia a 20 gauge intraarterial cannula was placed in to left radial artery and recorded 5 minute periods.

Anesthetic procedures and measured parameters were administered same ways except of PEEP levels.

All patients were received midazolam 2mg intravenously (IV) about five minute before induction. Anesthesia was induced with fentanyl( 1-3 mcgr/kg), propofol (2-3mg/kg), rocuronium (0,6 mg/kg). After intubation anesthesia was maintained with sevoflurane 2-3 % volume (to improve MAC 1 levels for sevoflorane). Remifentanyl was given continuously during surgery at a rate of 0.05-2 mcg/kg/min) (IV). Rocuronium was administered at a rate of 30 min time intervals during the anesthesia. Sugammadex was administered at the end of the surgery for reversing the neuromuscular blockage. Tramadol 1mg/kg, 40 mg meperidine and paracetamol 1g were administered for postoperative analgesia after trochars were removed. The concentration of volatile anesthetic was monitored with GE anesthesia machine. Patients were ventilated 6 lt/dk gas flow (50% oxygen with 50% air mixture). 6-8 ml/kg tidal volume, inspiration/ expiration rate 1/2 was maintained. Respiratory rate was 8-12 breaths. EtCO2 was kept within the range 35-45 mmHg. 5mmHg PEEP was administered in Group 5 PEEP, no PEEP was administered Group ZEEP. Fluid balance and blood replacement was maintained with %0.09 NaCl and ringer or colloid(Voluven Fresenius Kabi, Graz, Austria) solution IV. Body temperature was maintained normothermic by upper body forced air and warming pads. Laparoscopic pressure was maintained at below 14mmHg throughout the operation. Intraabdominal pressure was measured in mililitres of mercury through a Foley bladder catheter with 3 stopcocks connected to infusion set and pressure transducer. IT connected to the electronic monitor of anesthesia machine. (Datex -Ohmeda S/5 Compact, GE Healthcare, Finland) . After clamping the tube 100 ml Saline solution was injected in to the bladder. The transducer was replaced and zeroed to the urinary bladder level whenever the position changes throughout the procedure. Oscillation test was performed before started the IAP measurements. This measurements was performed into two position: basal, after induction, before insuflation, after insuflation, before desuflation, after desuflation values were measured in supine position; 30min, 45 min, 60min measurements in 30 degree reverse trendelenburg position (head of the bed elevated to 30 degree). Intraabdominal hypertension was defined as an IAP of 12 mmHg or higher, according to the consensus definations of the World Society for The Abdominal Compartment Syndrome.

After end of the operation all the anesthetic agents stopped and 4 mg/kg sugammadex was performed IV.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients
* planned sleeve gastrectomy procedures under general anesthesia
* ASA 2-3 status
* 18-60 years old

Exclusion Criteria:

* Documented coronary or periferal arterial disease,
* Unregulated diabetes mellitus,
* History of smoking,
* Symptoms of bowel or urinary bladder obstruction,
* Preoperative systolic pressure grater than 170 mmHg,
* Diastolic arterial pressure grater than 90mmHg,
* Pregnancy,
* Anemia (haematocrit levels under %30),
* Symptoms of increased intracranial pressure,
* Significant stenosis of the carotid arteries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 morbidly obese patients which planned sleeve gastrectomy procedures under general anesthesia (ASA 2-3 status) were included in this study. Patients were devided into 2 groups which was ventileted with no positive end expiratory pressure(Group 5PEEP n=30), and 5 cmH2O positive and expiratory pressure (Group ZEEP n=30). All the patients were right hand dominate.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
cerebral oximeter | 3 hours
  To determine the effect of zero PEEP (ZEEP) and 5 mmHg positive end expiratory pressure (5PEEP) on cerebral oximeter levels in morbid obese patients whose undergoing laporoscopic sleeve gastrectomy.

SECONDARY OUTCOMES:
IAP changes on cerebral oxygen values | 3 hours
  Second outcome is to investigate the effect of intraabdominal pressure changes on cerebral oxygen values in LSG.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur S Şeker, Study Director — Duzce University Faculty of Medicine Anesthesiology and Intensive Care Depth, Duzce, Turkey; Yavuz Demiraran, Principal Investigator — Canakkale 18 Mart University, School of Medicine Department of Anesthesiology and Reanimation, Canakkale, Turkey; Ziya Salihoğlu, Principal Investigator — Istanbul University Cerrahpaşa Medical Faculty, Anesthesiology and Intensive Care Depth, Istanbul, Turkey; Tarık Umutoğlu, Principal Investigator — Bezmialem Vakif University, Faculty of Medicine, Anesthesiology and Intensive Care Depth, Istanbul, Turkey; İsmet Özaydın, Principal Investigator — Duzce University Faculty of Medicine General Surgery Depth, Duzce, Turkey; Sami Doğan, Principal Investigator — Duzce University Faculty of Medicine General Surgery Depth, Duzce, Turkey
Locations (1):
- Duzce Univercity Medical Fauculty, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MS, Bai SJ, Lee JR, Choi YD, Kim YJ, Choi SH. Increase in intracranial pressure during carbon dioxide pneumoperitoneum with steep trendelenburg positioning proven by ultrasonographic measurement of optic nerve sheath diameter. J Endourol. 2014 Jul;28(7):801-6. doi: 10.1089/end.2014.0019. Epub 2014 Mar 5. PMID 24517270
- [Background] Yi M, Leng Y, Bai Y, Yao G, Zhu X. The evaluation of the effect of body positioning on intra-abdominal pressure measurement and the effect of intra-abdominal pressure at different body positioning on organ function and prognosis in critically ill patients. J Crit Care. 2012 Apr;27(2):222.e1-6. doi: 10.1016/j.jcrc.2011.08.010. Epub 2011 Oct 26. PMID 22033056
- [Background] Sprung J, Whalley DG, Falcone T, Warner DO, Hubmayr RD, Hammel J. The impact of morbid obesity, pneumoperitoneum, and posture on respiratory system mechanics and oxygenation during laparoscopy. Anesth Analg. 2002 May;94(5):1345-50. doi: 10.1097/00000539-200205000-00056. PMID 11973218